CLINICAL TRIAL: NCT00498251
Title: Does Inhaled Salbutamol Prevent Lung Edema After Thoracic Surgery? A Randomized Controlled Study
Brief Title: Prevention of Lung Edema After Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CER03-160
Record Dates: First submitted 2007-07-06; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-06

CONDITIONS: Lung Injury, Acute; Thoracotomy; Anesthesia; Intensive Care, Surgical; Extravascular Lung Water
Keywords: lung injury, acute; thoracic surgical procedures; lung cancer; salbutamol
MeSH Terms: conditions — Acute Lung Injury; Lung Neoplasms | interventions — Ipratropium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: inhalation of salbutamol (5 mg)
Drug: ipratropium

SUMMARY:
Background :

Acute lung injury (ALI) occasionally occurs after pulmonary resection and carries a bad prognosis with a high mortality rate ranging from 20 to 100%.

Objectives :

1. to evaluate pre-, intra- and postoperative changes in hemodynamics, oxygenation indices as well as intra- and extravascular lung water using simple thermodilution technique and continuous arterial pressure analysis
2. to test the efficacy of inhaled beta2 -adrenergic agonist versus anticholinergic agents to reduce lung edema in patients undergoing thoracic surgery and in pigs subjected to lipolysacharide-induced ALI.

Design of the research protocol:

* Prospective controlled trial including surgical patients with high risk factors for ALI (n=60) allocated to receive inhaled drugs (randomised, double-blind, cross-over mode).
* Main measurements:

Intra-thoracic blood volume, intra- and extra-vascular lung water, hemodynamic parameters (CO, systolic arterial pressure/flow variations, dPmax, MAP, CVP), oxygenation indices (PaO2/FIO2), ventilatory parameters, clinical outcome data, histochemical and pathological data.

Glossary CO = cardiac output; dPmax = maximal arterial pressure slope; SAP-V = systolic arterial pressure variations; Flow-V = Flow variations; MAP = mean arterial pressure; CVP = central venous pressure; PaO2=arterial oxygen pressure; FIO2= oxygen inspiratory fraction

DETAILED DESCRIPTION:
Material and Methods Patient selection Consecutive patients who require elective lung resection for cancer at the University Hospital of Geneva will be screened for the presence of risk factors for postoperative ALI or hydrostatic lung edema: age > 60 yrs, history of chronic alcohol consumption (>60g/day), prior radiation or chemotherapy, cardiac insufficiency (left ventricular ejection fraction < 40%, or a history of past acute heart failure), coronary artery disease (history of myocardial infarct, Q wave on the ECG, positive stress test or coronary angiogram), recent pneumonia (within 6 weeks of hospital admission), reduced diffusion capacity for carbon monoxide (DLCO < 60% of predicted values) and predicted postoperative lung perfusion of < 55% of total lung perfusion. Patients with at least 3 risk factors for postoperative lung edema will be considered eligible for the study. Patients undergoing pneumonectomy or presenting with intracardiac shunts, valvular diseases or aortic abdominal aneurysm will all be excluded as these conditions preclude valid measurements of extravascular lung water volumes. In addition, chronic treatment with inhaled bronchodilators, a history of any adverse reaction to bronchodilators and liver or kidney insufficiencies will be considered exclusion criteria.

This randomized double blind, cross-over study has been approved by the local university hospital ethics committee and written informed consent has been obtained from all selected patients.

The same team of pneumonologists, thoracic surgeons and anesthesiologists/intensive care physicians will be involved in the perioperative medical management. In addition to history and clinical examination, a standardized preoperative assessment includes chest radiography, ECG, pulmonary function testing as well as computed tomography scans and positron emission tomographies of the chest, abdomen and brain. Quantitative lung perfusion/ventilation scanning, brain imaging, maximal aerobic capacity and myocardial stress testing will be performed when appropriate in intermediate-to-high risk surgical candidates.

Operative and anesthetic management Routinely, antimicrobial prophylaxis with cefazoline will be administered for 24 hours and an epidural catheter was inserted at the 4th-5th or at the 5th-6th vertebral interspace. Thoracic epidural anesthesia (TEA) will be initiated preoperatively with the administration of bupivacaïne 0.25% and continued postoperatively with a lower dosage (bupivacaine 0.1%) that was combined with opiates (fentanyl 2 mcg/ml).

Each patient will be equipped with a 4-French femoral artery catheter and an internal jugular venous line that will be connected to a pulse contour cardiac output monitor (PV2024L; Pulsion Medical Systems AG, Munich, Germany).

After anesthesia induction, a left sided double-lumen endotracheal tube will be inserted and pressure support ventilation will be adjusted to optimize gas exchanges and minimize lung hyperinflation with low tidal volume (5-6 ml/kg), high inspiratory oxygen fraction (50-80%) and positive end expiratory pressure levels (PEEP, 4-12 cm H2O). Periodically, lung recruitment maneuvers will also be performed to re-open alveolar collapsed areas. Anesthesia will be maintained by infusing propofol targeted to achieve bispectral electroencephalographic values between 40 and 60. Lung resection with systematic lymph node dissection will be performed through an anterolateral muscle-sparing thoracotomy.

During surgery, intravenous crystalloids (Ringer-lactate solution) will be infused at a rate of 2-3 ml/kg/h and blood losses will be compensated with colloids (poly(0-2-hydroxy-ethyl)amidon, HAES 6%) and with red blood cell concentrates if the hemoglobin levels decreased below 80-90 g/L. At the end of surgery, all patients will be extubated in the operating theater after reversing the residual neuromuscular blockade with anticholinesterase agents. An active physiotherapy program including incentive spirometry, deep diaphragmatic breathing exercises and mobilization will be started in the high-dependency care unit (HDU). A maximal fluid balance of 500 ml per day will be targeted during the first 48 hours after surgery, by limiting fluid intakes including i.v. crystalloids (glucose-saline 0.45% 1 ml/kg/h), i.v. colloids (1/1 compensation of fluid losses through thoracic drains and oral beverages (500 ml on the day of surgery and 1'000-1'200 ml over the next two days).

Study design Within the first 36 hours after surgery, patients will received in random order nebulized salbutamol and nebulized ipratropium bromide at 4 consecutive sessions conducted at least 6 hours apart (figure 1). The treatment order will be generated from random number tables by an independent observer and concealed in sealed envelopes. The investigators, attending physicians and nurses will be blinded to the treatment group.

Over 10 minutes, either salbutamol (5 mg diluted in 5 ml normal saline) or ipratropium bromide (0.5 mg diluted in 5 ml normal saline) will be administered via a Cirrus nebulizer and a compressor (Wokingham, UK).

Measurements In addition to arterial blood sampling, complete sets of hemodynamic measurements will be performed as shown in figure 1: (a) preoperatively, before and 30 min after initiation of TEA, (b) 2 and 8 hours after surgery (postoperative day 0, [POD0]), before and 30 min after administration of salbutamol or ipratropium (6 hours apart in random order), (c) on the morning of the first postoperative day (POD1) on two consecutive sessions (6 hours apart in random order), before and 30 min after administration of salbutamol or ipratropium bromide.

Cardiac output (CO) and volumetric pulmonary variables will be obtained by the simple transpulmonary indicator dilution technique. Three consecutive measurements with less than 10% variations will be averaged. A fifteen milliliters bolus of 0.9% saline at 4°C will be injected through the central venous catheter into the right atrium and the change in temperature will be measured with the femoral artery thermistor tipped catheter. Using the mean transit time methods, intrathoracic blood volume, extravascular lung water and global end-diastolic volume will be calculated and indexed for the patient body weight (ITBVI, EVLWI and GEDVI, respectively). Heart rate (HR), stroke volume (SV) and maximal change in arterial pressure will be determined by beat-to-beat analysis of the arterial pressure wave. The systemic vascular resistance index (SVRI) will be calculated using standard formula. The ratio of EVLWI to ITBVI will be calculated as an index reflecting the permeability of the alveolar-capillary barrier.

Arterial oxygen pressure (PaO2 in mmHg) will be measured using a blood gas analyzer (ABL-510 analyzer, Radiometer, Copenhagen, Denmark) and will be related to the inspiratory O2 fraction to express the oxygenation index (PaO2/FIO2). In addition, chest radiograph scores (number of quadrants with >50% involvement with an alveolar filling process) will be recorded on POD0 (arrival in HDU) and POD1 (end of the study).

Outcomes The primary outcome measure will be a reduction in EVLWI within the first 24 hours after lung surgery. Secondary outcomes will be the PaO2/FIO2 ratio, hemodynamic data and radiological lung injury score.

Statistical analysis A sample size of 20 subjects provides the power (80%) to detect a 20% difference in EVLWI for a two-sided significance level of  = 0.05; in a preliminary study, we found a mean value of 9.1 ml/kg for EVLWI with a standard deviation (SD) of 2.2 ml/kg.

Results will be reported as M(SD), median (interquartile) or numbers (percentages). A p value of < 0.05 was considered significant in all analyses. All data will be analyzed with the SPSS statistical software (version 9.0, SPP, Chicago, IL). ANOVA for repeated measurements will be used to compare baseline values (preoperative, POD0 and POD1) followed by Bonferroni post-hoc tests. Paired and unpaired Student t tests will be used to assess and to compare the effects of bronchodilators. Furthermore, the correlation between changes in EVLWI, CI, ITBVI and PaO2/FIO2 will be analyzed by linear regression.

ELIGIBILITY:
Inclusion Criteria:

Patients with at least 3 risk factors for postoperative lung edema

* age > 60 yrs
* history of chronic alcohol consumption (>60g/day)
* prior radiation or chemotherapy
* cardiac insufficiency (left ventricular ejection fraction < 40%, or a history of past acute heart failure)
* coronary artery disease (history of myocardial infarct, Q wave on the ECG, positive stress test or coronary angiogram)
* recent pneumonia (within 6 weeks of hospital admission)
* reduced diffusion capacity for carbon monoxide (DLCO < 60% of predicted values)
* predicted postoperative lung perfusion of < 55% of total lung perfusion

Exclusion Criteria:

* pneumonectomy
* intracardiac shunts
* valvular diseases
* aortic abdominal aneurysm
* chronic treatment with inhaled bronchodilators
* a history of any adverse reaction to bronchodilators
* liver or kidney insufficiencies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
reduction in extravascular lung water | within the first 24 hours after lung surgery

SECONDARY OUTCOMES:
changes in oxygenation indices, hemodynamics and radiological lung injury score | within the first 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Ellenberger, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Licker M, Tschopp JM, Robert J, Frey JG, Diaper J, Ellenberger C. Aerosolized salbutamol accelerates the resolution of pulmonary edema after lung resection. Chest. 2008 Apr;133(4):845-52. doi: 10.1378/chest.07-1710. Epub 2007 Nov 7. PMID 17989152